CLINICAL TRIAL: NCT03239379
Title: A Multiple-Dose Study of Intravenous BNZ132-1-40 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioniz Therapeutics (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BNZ1-CT-102
Record Dates: First submitted 2017-07-31; First posted 2017-08-04 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Safety and Tolerability in Healthy Subjects
Keywords: cytokine inhibitor; IL-2; IL-9; IL-15

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo
- BNZ132-1-40 (Experimental): PEGylated BNZ-1 for Injection
  Interventions: Drug: BNZ132-1-40

INTERVENTIONS:
Drug: BNZ132-1-40 — Injectable peptide antagonist of IL-2, IL-9 and IL-15
  Other Names: BNZ-1
  Arms: BNZ132-1-40
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
This study is a single-center, randomized, single-blind, placebo (PBO)-controlled, multiple-dose study to characterize the safety, tolerability, PK, and PD of IV BNZ-1 administered to healthy adult subjects once weekly (QW) for 4 doses or once every other week (QOW) for 3 doses. Five cohorts of 6 subjects randomized 5 BNZ-1:1 PBO are planned to be enrolled in the trial. Participants will be followed for 4 weeks after the last dose for safety monitoring, and collection of PK and PD samples.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker.
2. Weight ≤100 kg (due to drug supply limitations).
3. Body Mass Index (BMI) ≥19 and <35 kg/m2.
4. Healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital signs (pulse rate, blood pressure, respiratory rate), and ECG.
5. Willing and able to consent and participate in the study.
6. Subject agrees not to receive any other investigational product or therapy while participating in this study.
7. Agrees to use adequate effective birth control methods prior to, during and for 30 days after the study.

Exclusion Criteria:

1. Clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study in the opinion of the Investigator.
2. History of cancer (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved).
3. History of or currently active primary or secondary immunodeficiency.
4. Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including tuberculosis [TB] or atypical mycobacterial disease [but excluding fungal infection of nail beds, minor upper respiratory tract infection, and minor skin conditions]), or any major episode of infection that required hospitalization or treatment with IV antibiotics within 30 days of screening or oral antibiotics within 14 days prior to screening.
5. Subject has received other investigational products or therapy in the past 30 days prior to study drug administration.
6. Serologic evidence of human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
7. Subject has received an immunization within 14 days prior to study drug administration.
8. History of alcohol or drug abuse within 1 year prior to screening.
9. Subject requires the ongoing use of prescription medication other than oral contraceptives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of treatment-emergent adverse events | 8 weeks
  general safety evaluation by principal investigator

SECONDARY OUTCOMES:
single-dose and steady state Cmax | 8 weeks
  plasma concentrations collected at multiple times after the first and last doses
single-dose and steady state AUC0-t | 8 weeks
  plasma concentrations collected at multiple times after the first and last doses
Steady-state Elimination half-life (t1/2) | 8 weeks
  plasma concentrations collected at multiple times after the last dose
Change from baseline for Regulatory T-cells (Tregs) | 8 weeks
  Flow cytometry of PBMCs at multiple time points post dose
Change from baseline for Natural Killer Cells | 8 weeks
  Flow cytometry of PBMCs at multiple time points post dose
Change from baseline for CD8+ central memory T-cells (Tcm) | 8 weeks
  Flow cytometry of PBMCs at multiple time points post dose

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Frohna, MD, PhD, Study Director — Bioniz Therapeutics, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No